CLINICAL TRIAL: NCT01279824
Title: A Randomized Controlled Trial of NMES vs. Traditional Dysphagia Therapy After Stroke
Brief Title: Adjunctive Neuromuscular Electrical Stimulation for the Rehabilitation of Swallowing
Acronym: ANSRS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Medical Rehabilitation Research (NCMRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: R21HD054752 (NIH); R21HD054752 (NIH)
Record Dates: First submitted 2011-01-07; First posted 2011-01-19 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Dysphagia
Keywords: swallowing, treatment, stroke,rehabilitation
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (Active Comparator): Patients will receive behavioral swallowing therapy comprising combination's of treatment strategies / exercises chosen from an approved hierarchy. This formulation of treatment will be designed and applied by the treating clinician.The treatment will be provided daily for a one-hour over a consecutive 3-week period.
  Interventions: Behavioral: swallowing therapy
- sham NMES (Placebo Comparator): Patients will receive behavioral swallowing therapy comprising combinations of treatment strategies / exercises chosen from an approved hierarchy with the addition of non stimulating electrodes. A faux NMES device will be utilized with an active current display and non stimulating electrodes. The treatment will be provided daily for a one-hour over a consecutive 3-week period.
  Interventions: Behavioral: swallowing therapy
- NMES therapy (Experimental): Patients will receive a protocol of standardized behavioral swallowing intervention combined with NMES. This formulation of treatment will be prescribed from a standard protocol and will be applied daily for one-hour over a consecutive 3-week period.
  Interventions: Behavioral: swallowing therapy

INTERVENTIONS:
Behavioral: swallowing therapy — Standardized behavioral swallowing intervention

SUMMARY:
Neuromuscular Electrical stimulation (NMES) for swallowing has recently been proposed for the treatment of dysphagia post stroke and is clinically receiving favor as a treatment modality, in the absence of strong research support. This study aims to investigate the effect of NMES therapy for dysphagia upon recovery of swallowing function following stroke. The study will follow a pilot randomized controlled trial design. Fifty one patients admitted to a sub-acute rehabilitation facility will be clinically screened for dysphagia, and randomized into one of three groups, NMES, sham NMES or usual care -behavioral swallowing therapy arm. All patients will be treated for one hour per day for 3 weeks, and their progress and outcome will be monitored. The results will add to the preliminary data on the effectiveness of this form of swallowing treatment for patients following stroke, and has the potential to enable more efficient allocation of resources to post-acute rehabilitation and thus benefit afforded to stroke patients, and the community.

DETAILED DESCRIPTION:
This pilot randomized controlled trial (N=51) includes stroke patients admitted to a sub-acute rehabilitation facility. Subjects will be clinically screened for dysphagia, and randomized into three groups, NMES, sham NMES or usual care -behavioral swallowing therapy arm. Following randomization, all subjects will undergo a video-x-ray (modified barium swallow) of swallowing to confirm the presence of oropharyngeal dysphagia and provide objective data about the nature and degree of dysphagia. All patients will be treated for one hour per day for 3 weeks, and their progress and outcome will be recorded. Participants will be independently evaluated by a blinded assessor at baseline, post treatment and at 3 months following treatment. The primary outcome will be improvement in clinical swallowing ability, oral intake level, and body weight. The results will add to the preliminary data on the effectiveness of this form of swallowing treatment for patients following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke identified by neurological and radiological examination
* Oropharyngeal dysphagia as confirmed by clinical and radiological examination
* No prior history of oropharyngeal dysphagia by patient and/or caregiver report
* No previous head/neck surgery or trauma that may impact swallowing ability
* No other/concomitant neurological disorders (e.g. Parkinson's disease) that would impact oropharyngeal swallowing ability. This does not include post-stroke deficits.
* Physician and patient/family agreement to participate.

Exclusion Criteria:

* Exposed to previous behavioral or NMES swallowing therapy within 6 months of admission
* Presence of progressive neurological disorder, such as ALS; Parkinson's or other neurologic disorders within the last 6 months;
* History of neurosurgery (either ablative or stimulatory), encephalitis or significant head trauma.
* History of a significant medical condition such as heart, liver, or renal disease; history or evidence of malignancy within the past 5 years other than excised basal cell carcinoma.
* Because of FDA Warnings, patients with cardiac demand pace makers will be excluded.
* Patients with evidence of significant cognitive impairment or dementia as reflected in a Mini-Mental test less than 23 and/or a score of 50% or less on the comprehension quotient on the Western Aphasia Battery.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Clinical response | 3 weeks post treatment
  Mann Assessment of Swallowing Ability (M.A.S.A)and Functional Oral Intake Scale (F.O.I.S) change, without significant weight loss or dysphagia-related complication
Full clinical response | 3 months post treatment
  Mann Assessment of Swallowing Ability (M.A.S.A)and Functional Oral Intake Scale (F.O.I.S) change, without significant weight loss or dysphagia-related complication.

SECONDARY OUTCOMES:
Recovery of pre-stroke diet | Baseline, 3 weeks (post treatment) and 3 months post
  comparison of diet intake
Dysphagia-related medical complications | Baseline,3 weeks ( post treatment) and 3 months post
  Occurance of chest infection, dehydration or significant weight loss
Biomechanic evaluation of swallowing function | Baseline and 3 weeks (post treatment)
  Modified barium swallow measurement will be used to document changes in swallowing biomechanics associated with change in swallowing following treatment.
Functional stroke recovery | Baseline, 3 weeks (post treatment) and at 3-months post treatment
  Modified Rankin Scale and the Modified Barthel Index will be used to measure functional stroke recovery.
Neurological status/Stroke severity | baseline, 3 weeks (post treatment) and at the 3-month post treatment
  National Institutes of Health Stroke Scale will be used to measure neurological status change.
Patient perception of swallowing ability | baseline, 3 weeks (post treatment) and at 3-months post treatment
  Using a visual analogue scale patients will indicate ability to swallow.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Carnaby-Mann, PhD, Principal Investigator — University of Florida
Locations (1):
- Siskin Hospital for Physical Rehabilitation, Chattanooga, Tennessee, United States

REFERENCES:
- [Background] Carnaby-Mann GD, Crary MA. Adjunctive neuromuscular electrical stimulation for treatment-refractory dysphagia. Ann Otol Rhinol Laryngol. 2008 Apr;117(4):279-87. doi: 10.1177/000348940811700407. PMID 18478837
- [Background] Carnaby-Mann GD, Crary MA. Examining the evidence on neuromuscular electrical stimulation for swallowing: a meta-analysis. Arch Otolaryngol Head Neck Surg. 2007 Jun;133(6):564-71. doi: 10.1001/archotol.133.6.564. PMID 17576907
- [Background] Carnaby-Mann GD, Crary MA. McNeill dysphagia therapy program: a case-control study. Arch Phys Med Rehabil. 2010 May;91(5):743-9. doi: 10.1016/j.apmr.2010.01.013. PMID 20434612